CLINICAL TRIAL: NCT04977284
Title: Noninvasive Neuroprosthesis for Autonomic Recovery After Spinal Cord Injury
Brief Title: Noninvasive Neuroprosthesis for Autonomic Recovery After SCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Praxis Spinal Cord Institute (Other); St. Paul's Hospital (Unknown)
Responsible Party: Principal Investigator, Andrei Krassioukov, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H21-00781
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCSCS (Experimental)
  Interventions: Device: DS7R, Digitimer, UK

INTERVENTIONS:
Device: DS7R, Digitimer, UK — Non-surgical spinal cord stimulation will be applied and electrical activity of muscles will be recorded.

SUMMARY:
This research study is being conducted to help explore the effects of non-invasive (non-surgical) spinal cord stimulation via sticky electrodes over the skin (transcutaneous spinal cord stimulation; TCSCS) on bowel, bladder and sexual function following spinal cord injury. Our primary aim is to determine the specific location and timing of TCSCS at various spinal cord levels in order to target bladder and bowel control (Study 1 and 2), and to assess the safety and effectiveness of TCSCS during bladder and bowel function assessments (Study 2 only). Participants may choose to participate in either Study 1 or 2.

ELIGIBILITY:
Inclusion Criteria:

* Resident of British Columbia, Canada with active provincial medical services plan
* Male or female, 18-65 years of age
* Chronic traumatic SCI (non-progressive, with complete motor paralysis) at or above the T10 spinal segment.
* >1-year post injury, at least 6 months from any spinal surgery.
* American Spinal Injury Association Impairment Scale (AIS) A, B.
* Willing and able to comply with all clinic visits and study-related procedures.
* Able to understand and complete study-related questionnaires (must be able to understand and speak English or have access to an appropriate interpreter as judged by the investigator).
* No painful musculoskeletal dysfunction, unhealed fracture, pressure sore, or active infection that may interfere with testing activities.
* Stable management of spinal cord related clinical issues (i.e., spasticity management).
* Women of childbearing potential must not be intending to become pregnant, currently pregnant, or lactating. The following conditions apply:

  1. Women of childbearing potential must have a confirmed negative pregnancy test prior to the baseline visit. During the trial, all women of childbearing potential will undergo urine pregnancy tests at their monthly clinic visits as outlined in the schedule of events.
  2. Women of childbearing potential must agree to use adequate contraception during the period of the trial and for at least 28 days after completion of treatment. Effective contraception includes abstinence.
* Sexually active males with female partners of childbearing potential must agree to use effective contraception during the period of the trial and for at least 28 days after completion of treatment.
* Must provide informed consent.

Exclusion Criteria:

* Presence of severe acute medical issue that in the investigator's judgement would adversely affect the participant's participation in the study. Examples include, but are not limited to clinically significant renal or hepatic disease; acute urinary tract infections; pressure sores; active heterotopic ossification; newly changed antidepressant medications [tricyclics]; or unstable diabetes.
* Recent treatment with OnabotulinumtoxinA into the detrusor muscle (relative contraindication).
* Ventilator dependent
* Use of any medication or treatment that in the opinion of the investigator indicates that it is not in the best interest of the participant to participate in this study.
* Intrathecal baclofen pump.
* Cardiovascular, respiratory, bladder, or renal disease unrelated to SCI or presence of hydronephrosis or presence of obstructive renal stones.
* Any implanted metal in trunk or spinal cord under the sites of application of electrodes (between anode and cathode).
* Participant is a member of the investigational team or his /her immediate family.
* Participant has undergone electrode implantation surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Activation of spinal circuits | Week 1
  Activation of spinal circuits is measured by the presence of motor evoked potentials or free run surface electromyography (EMG signal above baseline recorded from above muscles in response to TCSCS applied between spinous processes T10-11, T11-12, T12-L1, and L1-L2 (conus medullaris).

SECONDARY OUTCOMES:
Safety and efficacy during Urodynamic Testing (UDS) | Week 2 to 4
  Safety and efficacy of UDS is measured by presence of detrusor contractions (voiding function) while relaxing the EUS, i.e. to avoid detrusor sphincter dyssynergia and independently enhance EUS tone (storage function) without adverse cardiovascular effects.
Safety and efficacy during Anorectal Manometry (ARM) | Week 2 to 4
  Safety and efficacy of ARM is measured by presence of an immediate increase in anorectal pressure without adverse cardiovascular effects.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Krassioukov, MD, PhD, Principal Investigator — University of British Columbia

IPD SHARING:
Plan to Share IPD: No